CLINICAL TRIAL: NCT06397612
Title: Registry on the Short- and Medium-term Efficacy of Low-dose Peripheral Nerve Stimulation of the Pudendal Nerve in Patients With Pudendal Nerve in Patients With Erectile Dysfunction
Brief Title: Efficacy of Low-dose Percutaneous Electrical Stimulation in Patients With Erectile Dysfunction.
Acronym: Low-NEEP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Camilo Jose Cela University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Low-NEEP
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Pudendal Nerve Injury; Erectile Dysfunction; Electric Stimulation
Keywords: Erectile Dysfunction; Percutaneous Electrical Neurostimulation; Low Dose; Pudendal Nerve
MeSH Terms: conditions — Erectile Dysfunction | interventions — Contraceptives, Oral

STUDY DESIGN:
Intervention Model Description: The study corresponds to a non-randomized, single treatment arm, prospective, multicenter study. The subject, the assignor, the physiotherapist, the statistician and a person in charge of activating the protocol will know the stimulation parameters, to adjust, monitor and apply the treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group I (Experimental): The intervention protocol for Group I peripheral nerve electrostimulation will have the following parameters:
  Patients will be intervened with stimulation continuously, at a frequency of 20 Hertz, a pulse width of 200 µs and for a total of 20 minutes. The intensity will be set at the maximum tolerated by the patient.
  Interventions: Other: Low Dose

INTERVENTIONS:
Other: Low Dose — Patients will be intervened with stimulation continuously, at a frequency of 20 Hertz, a pulse width of 200 µs and for a total of 20 minutes. The intensity will be set at the maximum tolerated by the patient.

SUMMARY:
Erectile dysfunction is known as any alteration that produces a modification in the erectile response, whether it is due to organic, psychogenic or relational causes. Peripheral percutaneous nerve stimulation is performed using a needle to stimulate the peripheral nerves in such a way as to stimulate most of the area of the structure, stimulating sensory and motor nerve endings in the deeper tissues.

DETAILED DESCRIPTION:
Patients will undergo continuous stimulation at a frequency of 20 Hertz, a pulse width of 200 µs and for a total of 20 minutes. The intensity will be set at the maximum tolerated by the patient, observing significant changes in erectile function after transanal stimulation at intensities between 20 and 100 mA.

ELIGIBILITY:
Inclusion Criteria:

Males Ages between 18-60 years old

Primarily organic cause diagnosed by Doppler:

* Peak-systolic velocities (PSV).
* Tele-diastolic velocity (DTV).
* Resistance Index (RI) Patients with ≤ 6 months since first assessment. Initial IIEF-EF questionnaire scores: 11-25 points. (mild to moderate erectile dysfunction) Active sexual life (more than 4 attempts per month).

Exclusion Criteria:

Pelvic surgeries History of Peyronie's disease Penile surgeries, except circumcision or frenuloplasty Priapism Pelvic radiation Female

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 24 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
International Index of Erectile Function (IIEF-EF) | 4 months
  It is an index that assesses erectile function in a purely subjective way. It is the most recognized and used, and consists of six questions in which the frequency and firmness of the erection, the capacity of penetration, the capacity and frequency of maintenance and the confidence in the erection are evaluated. According to the questionnaire, dysfunction is classified as: no ED (26-30 points), mild (22-25 points), mild to moderate (17-21 points), moderate (11-16 points) and very strong (6-10 points). A score equal to or greater than 4 points will be considered a significant change. Measurement pre, one week after the intervention, one month after the intervention, three months after the intervention.
Erection Hardness Scale (EHS) | 4 months
  The following will be considered significant changes men who improved by more than 3 points what in the initial phase was below a score of 2 points. The questionnaire score depends on the rating of erection hardness according to the following parameters: 0 (penis does not enlarge); 1 (penis is larger, but not hard); 2 (penis is hard but not hard enough for penetration); 3 (penis is hard enough to penetrate, but not completely hard); and 4 (penis is completely hard and rigid). Measurement pre, one week after the intervention, one month after the intervention, three months after the intervention.
Premature Ejaculation Diagnostic Tool (PEDT) | 4 months
  Helps identify patients who may be suffering from premature ejaculation. Measurement pre, one week after the intervention, one month after the intervention, three months after the intervention.
Quality of Life Scale | 4 months
  It is used to subjectively assess the patient's opinion of his or her quality of life, based on 4 main aspects: physical, psychological, social and environmental health.Measurement pre, one week after the intervention, one month after the intervention, three months after the intervention. The scale is measured by 26 items, divided into 4 dimensions. Each dimension is independent. The higher the score, the higher the patient's quality of life.
Self-Esteem And Relationship Questionnaire (Sear) | 4 months
  A questionnaire used for research and/or clinical practice use on self-esteem, in this case for patients with erectile dysfunction. Measurement pre, one week after the intervention, one month after the intervention, three months after the intervention. The scale is measured from 0 to 100 points, with 0 being the worst score and 100 being the best.

CONTACTS AND LOCATIONS:
Overall Officials: Álvaro Navas Mosqueda, Principal Investigator — Camilo Jose Cela Univerity
Locations (1):
- LYX Instituto de Urología, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yafi FA, Jenkins L, Albersen M, Corona G, Isidori AM, Goldfarb S, Maggi M, Nelson CJ, Parish S, Salonia A, Tan R, Mulhall JP, Hellstrom WJ. Erectile dysfunction. Nat Rev Dis Primers. 2016 Feb 4;2:16003. doi: 10.1038/nrdp.2016.3. PMID 27188339
- [Background] Beltra P, Ruiz-Del-Portal I, Ortega FJ, Valdesuso R, Delicado-Miralles M, Velasco E. Sensorimotor effects of plasticity-inducing percutaneous peripheral nerve stimulation protocols: a blinded, randomized clinical trial. Eur J Pain. 2022 May;26(5):1039-1055. doi: 10.1002/ejp.1928. Epub 2022 Mar 3. PMID 35191131
- [Background] Peters KM, Carrico DJ, Perez-Marrero RA, Khan AU, Wooldridge LS, Davis GL, Macdiarmid SA. Randomized trial of percutaneous tibial nerve stimulation versus Sham efficacy in the treatment of overactive bladder syndrome: results from the SUmiT trial. J Urol. 2010 Apr;183(4):1438-43. doi: 10.1016/j.juro.2009.12.036. Epub 2010 Feb 20. PMID 20171677